CLINICAL TRIAL: NCT01407263
Title: A Randomized Trial of Modifications to Radical Prostatectomy
Brief Title: Trial of Modifications to Radical Prostatectomy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 11-096
Record Dates: First submitted 2011-07-29; First posted 2011-08-02 (Estimated); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
Keywords: radical prostatectomy; anastomotic suturing; lymph node dissection; 11-096
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Antibiotic Prophylaxis; Hemostasis

ARMS (4):
- Lymphadenectomy vs. no lymphadenectomy (Experimental): In patients randomized to standard, only the nodal packet under the external iliac vein and above the obturator nerve will be dissected. For patients randomized to the modified template, the external iliac, hypogastric and obturator fossa nodal groups will be removed.No lymph nodes will be removed in patients randomized to the no PLND arm.
  Interventions: Procedure: Lymph node template
- Transverse versus vertical closure of the port site incision (Closed as of 9/30/2021) (Experimental)
  Interventions: Procedure: Transverse versus vertical closure
- One vs. three days of antibiotic prophylaxis (Closed as of 9/30/2021) (Experimental)
  Interventions: Drug: antibiotic prophylaxis
- Hemostatic agent vs. no hemostatic agent (Experimental)
  Interventions: Drug: Hemostatic Agent

INTERVENTIONS:
Procedure: Lymph node template — Inclusion of the external iliac, hypogastric and obturator fossa nodal groups in the template undergoing a Radical Prostatectomy. Modifying the template for lymph node dissection may lead to removal of additional affected nodes, reducing the chance of recurrence. .No lymph nodes will be removed in patients randomized to the no PLND arm.
  Arms: Lymphadenectomy vs. no lymphadenectomy
Procedure: Transverse versus vertical closure — Transverse versus vertical closure of the port site incision
  Arms: Transverse versus vertical closure of the port site incision (Closed as of 9/30/2021)
Drug: antibiotic prophylaxis — One vs. three days of antibiotic prophylaxis at catheter removal
  Arms: One vs. three days of antibiotic prophylaxis (Closed as of 9/30/2021)
Drug: Hemostatic Agent — For the patients randomized to routine indwelling HA agent use, the operating surgeon may choose to use either Surgicel™, Surgicel SNoW™, Arista™, FloSeal or surgeon's choice HA directed at the prostatic fossa, ligated dorsal vein complex, or neurovascular bundles. Because there is no standard HA or method of application, the surgeon will apply the HA according to the surgeon's experience and document both the HA used, and the location applied in the operative report. For patients randomized to no routine indwelling HA use, surgeons will only apply a HA if they are unable to achieve hemostasis using traditional means or feel it would be unsafe to complete the operation without using a HA for additional hemostasis. Providers in either arm may use HA as needed provided the intention is not to leave the HA indwelling.
  Arms: Hemostatic agent vs. no hemostatic agent

SUMMARY:
This trial will evaluate whether the following aspect of surgical technique influence outcome: Lymph node dissection. In some patients, scans taken before surgery show that a lymph node has cancer. Surgeons make sure to remove those affect lymph nodes and all other lymph nodes in the area. However, it is not known whether removing lymph nodes helps prostate cancer patients whose scans do not show positive nodes. In this study, patients with clear scans will either receive a lymph node dissection or not."

ELIGIBILITY:
Inclusion Criteria:

* Patients do not have to be eligible for both modifications to be included in the study.

Lymphadenectomy vs no lymphadenectomy:

* Patients 21 years or older scheduled for radical prostatectomy for treatment of prostate cancer with one of the consenting surgeons at MSKCC

Hemostatic agent vs. no hemostatic agent

* Patients 21 years or older scheduled for minimally invasive radical prostatectomy for the treatment of prostate cancer with one of the consenting surgeons at MSKC

Exclusion Criteria:

Lymphadenectomy vs no lymphadenectomy

* Presence of positive/suspicious pelvic nodes on MRI, CT or PSMA scan (positive/suspicious defined as a pelvic node >15mm in short axis on CT or MRI, a PSMA avid node, or a node with abnormal morphology such as roundness or irregularity or loss of fatty hilum)
* Any prior pelvic radiation therapy used to treat prostate cancer

Hemostatic agent vs. no hemostatic agent

* No additional exclusion criteria

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3204 (Actual)
Dates: Start 2011-07; Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Patient-reported hernia | 1 year
  Patient-reported hernia is a routine assessment on post-operative questionnaires completed by prostate cancer patients at MSKCC. The questionnaire asks about hernia near the surgical scar and if there has been a need for surgical repair of the hernia.

SECONDARY OUTCOMES:
To evaluate whether a modification to the template for lymph node dissection reduces biochemical recurrence rates | 2 years
  Biochemical recurrence is defined as any postoperative PSA of 0.2 ng / mL or higher, or treatment with hormones, radiotherapy or chemotherapy starting six months or more after radical prostatectomy.
urinary tract infection (UTI) | within 10 days
  urinary tract infection (UTI) within 10 days of catheter removal. We will use the CDC's definition of UTI: symptomatic UTI diagnosed in patients with positive urine cultures (≥100,000 microorganisms per cm3) and at least one of the following signs or symptoms with no other recognized cause: fever (>38oC), urgency, frequency, dysuria or suprapubic tenderness.50 UTI is routinely captured by clinical staff as a surgical complication.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Vickers, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan Kettering Cancer Center at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Bergen (Consent Only), Montvale, New Jersey
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center @ Nassau (Consent only), Uniondale, New York

REFERENCES:
- [Derived] Touijer KA, Vertosick EA, Sjoberg DD, Liso N, Nalavenkata S, Melao B, Laudone VP, Ehdaie B, Carver B, Eastham JA, Scardino PT, Vickers AJ. Pelvic Lymph Node Dissection in Prostate Cancer: Update from a Randomized Clinical Trial of Limited Versus Extended Dissection. Eur Urol. 2025 Feb;87(2):253-260. doi: 10.1016/j.eururo.2024.10.006. Epub 2024 Oct 29. PMID 39472200
- [Derived] Gaffney CD, Vertosick EA, Laudone V, Goh AC, Carlsson SV, Pietzak E, Donahue T, Smith R, Touijer K, Vickers AJ, Ehdaie B. Randomized Trial of Transverse vs Vertical Extraction Site Incision After Robotic Radical Prostatectomy. J Urol. 2024 Sep;212(3):401-408. doi: 10.1097/JU.0000000000004066. Epub 2024 Aug 8. PMID 39115122
- [Derived] Touijer KA, Sjoberg DD, Benfante N, Laudone VP, Ehdaie B, Eastham JA, Scardino PT, Vickers A. Limited versus Extended Pelvic Lymph Node Dissection for Prostate Cancer: A Randomized Clinical Trial. Eur Urol Oncol. 2021 Aug;4(4):532-539. doi: 10.1016/j.euo.2021.03.006. Epub 2021 Apr 15. PMID 33865797
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm